CLINICAL TRIAL: NCT04401332
Title: Integrating Patient-Reported Outcomes Into Routine Primary Care: Monitoring Asthma Between Visits
Brief Title: A Randomized Controlled Trial of AppS to Home Monitor Your Asthma
Acronym: ASTHMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-0038; 2018P002394 (Other: Mass General Brigham)
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: patient-reported outcomes (PROs); mobile health (mHealth) apps; asthma; electronic health record (EHR); health information technology; implementation research; mobile phone
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: mobile health app
- Usual Care (No Intervention)

INTERVENTIONS:
Other: mobile health app — asthma symptom monitoring via a clinically integrated mobile health (mHealth) app installed on patients' smartphones
  Arms: Intervention

SUMMARY:
The objective of this study is to design, implement, and evaluate the impact of an adapted health information technology(IT)-enabled practice model for asthma symptom monitoring using patient-reported outcomes (PROs) in a primary care setting. Adults over 18 years of age with asthma will be recruited at primary care clinics and randomized to either 1) asthma symptom monitoring via the mobile health (mHealth) app; or 2) usual care. The investigators will collect data on patient-reported asthma quality of life and asthma-related healthcare utilization. We will also study barriers and facilitators to implementation of the mHealth app and health IT-enabled practice model.

DETAILED DESCRIPTION:
The specific aims of this study are:

1. Adapt our existing health IT-enabled practice model for asthma symptom monitoring using PROs to a primary care population. The health IT-enabled practice model is comprised of the following: an mHealth app that can be installed on patients' smartphones that integrates into clinical workflow; and an asthma PRO dashboard in the electronic health record (EHR) for clinicians.
2. Implement the adapted health IT-enabled practice model in 7 primary care community clinics, identify a cohort of eligible asthma patients to participate, and train clinicians and clinical staff.
3. Rigorously evaluate the impact of this new health IT-enabled practice model using a randomized controlled trial study in which we enroll 500 asthma patients (250 intervention, 250 usual care) by primary care clinician. We will measure patient-reported asthma quality of life and asthma-related healthcare utilization (defined as urgent care and emergency room visits and hospitalizations) as our primary and secondary outcomes, respectively. We will use mixed methods to identify barriers and facilitators to implementation and factors that affect sustainable spread and scale as per the Non-adoption, Abandonment, Scale-up, Spread, and Sustainability (NASSS) framework.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking
* 18 years of age
* Regularly uses (most days) a compatible smartphone (iOS or Android)
* Able to provide consent
* Seen for primary care within the last 12 months at one of the 7 outpatient primary care clinics that are part of the Brigham & Women's Hospital (BWH)/ Brigham & Women's Faulkner Hospital (BWFH) practice-based research network.
* At least one visit coded for asthma within 12 months prior to screening, including inpatient, emergency department, urgent care/walk-in, and specialist visits.

Exclusion Criteria:

* Deemed inappropriate for study, per judgment of the BWH/ BWFH primary care provider
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Asthma-related patient-reported quality of life | 6 months from enrollment
  Asthma-related patient-reported quality of life assessed using the 15-item Mini Asthma Quality of life Questionnaire (AQLQ)
Asthma-related patient-reported quality of life | 12 months from enrollment
  Asthma-related patient-reported quality of life assessed using the 15-item Mini Asthma Quality of life Questionnaire (AQLQ)

SECONDARY OUTCOMES:
Asthma-related healthcare utilization | 12 months from enrollment
  Asthma-related healthcare utilization, defined as number of urgent care and emergency room visits, and number of hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Rudin, PhD, Principal Investigator — RAND; Anuj K Dalal, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Rudin RS, Plombon S, Sulca Flores J, Sousa JL, Rodriguez J, Foer D, Lipsitz S, Edelen MO, Bates DW, Arcia A, Dalal AK. Between-Visit Asthma Symptom Monitoring With a Scalable Digital Intervention: A Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e256219. doi: 10.1001/jamanetworkopen.2025.6219. PMID 40266619